CLINICAL TRIAL: NCT06928597
Title: Global Postural Reeducation (GPR) in the Treatment of Patients With Non-Specific Chronic Low Back Pain: A Randomized Sham-Controlled Clinical Trial
Brief Title: Effects of GPR on Non-Specific Chronic Low Back Pain
Acronym: GPRSHAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, KAREN VALADARES TRIPPO, PhD, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FU_Bahia
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: Low back pain; Global Posture Reeducation; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (EG) - GPR (Experimental): The experimental group (EG) will receive GPR sessions. Participants will receive treatment through GPR postures in each session, regardless of the group. A minimum of one and a maximum of two postures will be chosen, what will be evolved progressively put node minimum 15 (fifteen) minutes, case two postures are chosen and, at most, 30 (thirty) minutes, in the case of only one posture. Both groups will be treated for 30 (thirty) minutes, once a week, for eight weeks, totaling eight sessions. One physiotherapist with complete training in the RPG method will carry out the EG services. For the EG, the guidelines for breathing during GPR will be rhythmic breathing, prioritizing the associated expiration and contraction of the abdominal muscles and of the floor pelvis during exhalation.
  Interventions: Procedure: Global Postural Reeducation; Procedure: Global Postural Reeducation Sham
- Control Group (CG) - GPR-SHAM (Sham Comparator): The Control Group (CG) will receive GPR-SHAM sessions. In each session, participants will receive treatment through GPR postures regardless of the group. A minimum of one and a maximum of two postures will be chosen, what will be evolved progressively put node minimum 15 (fifteen) minutes, case two postures are chosen and, at most, 30 (thirty) minutes, in the case of only one posture. Both groups will be treated for 30 (thirty) minutes, once a week, for eight weeks, totaling eight sessions. The participants should dress in bathing, light, or gym clothes to feel comfortable during the sessions. One physiotherapist will be trained to carry out the RPG-SHAM in the CG.
  The simulation of the method will be carried out with the withdrawal of two important elements of the original method: the technique of contraction-relaxation and the guidelines from the breathing rhythm with prioritization of expiration.
  Interventions: Procedure: Global Postural Reeducation; Procedure: Global Postural Reeducation Sham

INTERVENTIONS:
Procedure: Global Postural Reeducation — Global Postural Reeducation, better known as GPR, was developed by Philippe Souchard in the 1980s and involves a sequence of postures or treatment positions, including the main ones: frog on the ground with arms open; frog on the ground with arms closed; frog in the air with arms open; frog in the air with arms closed; standing against the wall; standing at the center; anterior tilt sitting; anterior tilt standing.
  GPR is based on the concept of proprioception and inhibition. Souchard (2016) describes RPG as a proprioceptive method of inhibition, where proprioception refers to the body's ability to perceive its position in space, and inhibition refers to the muscle relaxation induced after intense contraction. This principle is applied through the postures and techniques used in treatment, aiming to correct postural deviations, promote one bigger conscious body, and relieve pain.
  Other Names: GPR or Posture Reeducation
Procedure: Global Postural Reeducation Sham — Global Postural Reeducation Sham is the comparator group.
  Other Names: GPR-SHAM

SUMMARY:
Introduction: Low back pain affects approximately 18.5% of the Brazilian population in adulthood, significantly impacting the quality of life and generating substantial costs for the health system. The Global Postural Reeducation Method (GPR) is a promising therapeutic alternative due to its multidimensional approach, capable of improving postural control and reducing pain. Objectives: to evaluate the Efficacy of the RPG method compared to simulated RPG (SHAM) in treating patients with chronic nonspecific low back pain. Methods: Randomized sham-controlled clinical trial. Forty-two adult individuals with chronic nonspecific low back pain will be recruited and distributed into two groups: the Experimental Group (EG), which will receive GPR sessions, and the Control Group (CG), which will receive RPG-SHAM sessions. Both groups will be treated for 30 minutes once a week for 8 weeks. Descriptive analysis will be performed, continuous variables will be summarized to the mean, and standard deviation and categorical variables will be summarized as absolute and relative frequencies. To assess the effects of the intervention over team, analysis of variance (ANOVA) with repeated measures will be used, with a significance level of 5% (p < 0.05). Expected Results: This study is expected to provide robust evidence on the effectiveness of RPG in treating patients with low back pain, contributing to a better understanding of this complex health condition. The results will potentially positively impact the clinical practice of Orthopedic Physiotherapy, offering an exercise-based and accessible approach for treating patients with low back pain.

DETAILED DESCRIPTION:
Low back pain is the most prevalent musculoskeletal condition in the world. According to the Institute for Health Metrics and Evaluation (IHME), there are 570 million prevalent cases worldwide, accounting for 7.4% of the Years Lived with Disability (YLD) or Years Lived with Inability. Of these conditions, low back pain is the leading cause of disability in more than 160 countries. Given this, it is known that this condition significantly impacts quality of life and generates substantial costs for health systems worldwide. In Brazil, approximately 18.5% of the population in the adult phase complains of pain at some moment in life. Still in the country, a study showed that between 1990 and 2017 this condition increased by 26.83%, being one of the three most significant causes of Disability Adjusted Life Years (DALYS) or Years of Life Lost Adjusted for Disability.

Global Postural Reeducation (GPR) is one method of proprioceptive inhibition that can facilitate movement. It was developed by Phillippe Emanuel Souchard in 1987 and is based on the theory of myofascial chains. The method's premise is that a change that presents in a particular group of muscles resonates in compensations and alterations throughout the myofascial chain. Therefore, the technique aims to reorganize these changes.

These corrections are made through concentric isometric exercises with manual resistance imposed for the therapist carried out to the far away of one stretching progressive and sustained in order to inhibit hyperactivated muscles through a specific sequence of active postures in increasingly eccentric positions of the static muscles applied in joint de-coaptation also progressive. The postures do not have a relationship of dependence and are chosen after a specific evaluation of the method.

Some research has been developed using this method in the last few years. The object of study in these studies varies between the effects on the treatment of nonspecific postural deviations, neck pain, and back pain (nonspecific). There are even studies that compare the treatment of low back pain with other methods. However, most lack methodological rigor, and none are compared with the RPG-SHAM.

The World Health Organization (WHO) guideline for non-surgical treatment of chronic primary low back pain in adults in primary and community care settings, published in 2023, recommends physical exercise and manipulative therapy as indicated alternatives. Thus, in view of its characteristics, where it is used for exercises to stimulate the inhibition of the hypertonic muscles and the therapy manipulative applied during the execution, the method GPR can be one alternative therapy to the low back pain chronicle nonspecific. Furthermore, as healthcare professionals frequently recommend this method, it is essential to check your effectiveness one time when there is a lack of scientific evidence and the need for studies with more considerable rigor methodological, as comparing the method with one procedure identical but simulated ( SHAM ), that is a sham-controlled study.

Thus, knowing the effects of the GPR method in reducing chronic nonspecific low back pain can contribute to the clinical practice of the physiotherapist since it is a non-pharmacological intervention based on exercises and that is widely inserted and disseminated in physiotherapy services but with little research that supports evidence-based practice. There is, therefore, a lack of high-quality studies in the scientific literature that evaluate the effects of this procedure in the management of chronic nonspecific low back pain in comparison with a sham group to support its therapeutic indication. Given the above, this research aims to evaluate the effectiveness of the GPR method compared to GPR-SHAM in treating people with chronic nonspecific low back pain through a randomized, sham-controlled clinical trial.

JUSTIFICATION:

Low back pain is an apparent public health problem that contributes to worsening quality of life and overloading health services. It is also a potential employment problem that causes many economically active individuals to be removed from their work environments. Recent epidemiological studies have shown the high prevalence of this complex health condition, which reinforces the importance and need for a practical approach.

Several therapeutic approaches are recommended in the guidelines for the treatment of low back pain, such as those from NICE, JOSPT, and WHO. The recommended therapies are health education, manual therapy, and physical exercise. Although not mentioned in these documents, it consists of a proprioceptive method of muscle inhibition; that is, it is a physical therapy based on exercises.

Data available on the Souchard GPR Institute-SP website report that about 22.000 (twenty-two thousand) physiotherapists practice GPR in Brazil and more than 17 (seventeen) other countries. However, Evidence-Based Practice (EBP) still has many limitations since several available studies lack methodological rigor and have a high risk of bias and sometimes questionable results due to the lack of control in conducting the studies.

In a study of meta-analysis, "Effectiveness of Global Postural Reeducation in Chronic Nonspecific Low Back Pain: Systematic Review and Meta-Analysis" even after a careful and in-depth search in the databases, including also using from the literature gray, due to the very few studies available about the GPR method for the outcome of this research, showed that no research performed masking of the patients. In addition, the article also demonstrated that just four of the eight articles found had notes bigger than five after the assessment from the PEDro scale, with one getting a score of two.

Therefore, masking patients in clinical studies is a fundamental practice to control biases, and an effective way to carry out this masking is through a sham-controlled group. In that model, the group control receives one simulated intervention similar to the original one, allowing the real effect to be isolated from the therapy.

In a study which investigated the effects of dry cupping therapy compared to sham cupping therapy in the treatment of chronic nonspecific low back pain, it was possible to identify that there was no difference between the interventions, showing what if treats of one treatment ineffective. In this form, the search with one sham-controlled group was essential to verify the effectiveness of the intervention and contribute scientific information to decision-making by healthcare professionals.

Research with a more significant scientific quality contributes to professionals' health commitment to offering community treatments adequately tested, with known and evidence-based effects. Therefore, this research project aims to contribute to a more significant understanding of the treatment of people with low back pain chronicle nonspecific, in addition to having the possibility of promoting evidence for an accessible, non-pharmacological, and potentially effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 55 years with chronic non-specific low back pain,
* Participants who voluntarily agree to participate and sign the Free and Informed Consent Form,
* Participants who have never done any treatment with the GPR method, and
* Participants who have not been undergoing physiotherapy treatment for at least 2 months.

Exclusion Criteria:

* Patients with pain lumbar acute, or it is, with symptoms gifts there is less of dose weeks, what carried out blocking medicinal in the column us last six months;
* Patients with hernia of disk of type extruded and/or kidnapped;
* Patients in possess or be in investigation of any kind of neoplasia;
* Patients who have undergone any type of surgery with placement of any type of prosthesis in the spine;
* Intellectual or sensory disability that prevents them from understanding commands or describing symptoms;
* Patients who have a significant change in tactile sensitivity that prevents them from reporting any symptoms;
* Patients who have any type of vestibular changes;
* Serious pathologies of the spine;
* Amputation of upper or lower limbs;
* Spinal Cord Injury;
* Low back pain with sacroiliac irradiation; any type of rheumatic diseases, such as: Rheumatoid Arthritis, Fibromyalgia, and others;
* Patients that be performing or carried out last two months any type of conservative treatments, such as: Acupuncture, hydrotherapy, manual therapy, Pilates, conventional physiotherapy, and others; and
* Patients who have travel plans in the coming months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Gradiation | pre and post eight weeks of intervention.
  Pain will be assessed three times: at rest, after a short walk, and during stem flexion using the Scale Visual Analog (EVE). This scale consists of a graduated horizontal line from 0 to 10, where 0 (zero) represents absence of pain and 10 (ten) represents maximum unbearable pain. Higher scores mean greater pain intensity.

SECONDARY OUTCOMES:
Range of motion (ROM) of the spine (Adams test) | pre and post eight weeks of intervention.
  The Adams test will be used to assess the range of motion during the spine flexion. The physiotherapist will ask the patient to stand barefoot, with feet hip-width apart and knees extended. Then, the physiotherapist will request one flexion before the stem, keeping the legs extended and avoiding compensations while the head and your shoulders remain relaxed. If the patient cannot touch the floor with their hands, the distance from the middle finger to the floor will be measured and recorded using a standard tape measure. Greater ranges of motion mean greater mobility of the evaluated segment.
Range of motion (ROM) of the spine (Inclinometer) | pre and post eight weeks of intervention.
  This instrument measures the inclination of a body segment relative to gravity, providing accurate data on joint mobility. To measure trunk rotation, the physical therapist will place the inclinometer on the patient's sternum, asking them to rotate the trunk as much as possible to both sides while the pelvis remains fixed. In the assessment of trunk flexion, the inclinometer will be placed on the upper part of the sacrum, and the patient will be instructed to lean forward as much as possible, keeping the knees extended. The inclinometer will remain in the same position for spine extension, and the patient will be requested to lean back as much as possible. The readings of the angles in each one of these positions will be recorded and compared to assess a range of motion and identify potential limitations or asymmetries. Greater ranges of motion mean greater mobility of the evaluated segment.
Postural Organization (photogrammetry) | pre and post eight weeks of intervention.
  The photos will be registered in the views front anterior and posterior, right and left lateral, following specific anatomical references. To meet the research objectives, additional markings will be added to the vertebrae with a circular sticker of 19mm in diameter in the colors green, lemon, or pink: seventh cervical, first and seventh thoracic, fourth and fifth lumbar.
Activity and participation assessment - World Health Organization Disability Assessment Schedule (WHODAS 2.0) | pre and post eight weeks of intervention.
  Assessment Schedule (WHODAS 2.0) will be used to assess patients' activities and participation. This tool consists of 36 items grouped into six main domains: cognition, self-care, interpersonal relationships, daily living activities, and social participation (CASTRO et al., 2019). Scores range from 0 to 100, with higher scores indicating greater functional limitation. The WHODAS 2.0 score ranges from 0 to 40, where higher values indicate greater disability.
Lower limb strength (sit-to-stand test - SST) | pre and post eight weeks of intervention.
  The test will be performed with a standard-height chair firmly on the floor. The physical therapist will instruct the patient to stand up and sit down again on command. Test score ranges from 0 to 5, considering the moments of sitting and standing. The time for the task will be timed. The time taken to complete the test is the main measure. The faster the individual can stand up and sit down 5 times, the better the performance.
Functional mobility (TUG) Functional mobility - Timed Up and Go (TUG test). | pre and post eight weeks of intervention.
  This test measures the time it takes for the patient to stand up from a chair, walk three meters, navigate around an obstacle, and return to the chair. The patient will receive proper guidance from the physiotherapist, who will stand one meter away. Scoring is based on the time taken, with shorter times indicating better performance.
Quality of life - Short Form 36 Health Survey (SF36) | pre and post eight weeks of intervention.
  The Short Form 36 Health Survey (SF36)** is a validated questionnaire designed to assess quality of life. It consists of 36 questions grouped into eight distinct domains: functional capacity, physical limitations, pain, general health status, vitality, social aspects, emotional aspects, and mental health. Higher scores indicate better health.
Anxiety and depression - Hospital Anxiety and Depression Scale (HAD) | pre and post eight weeks of intervention.
  To evaluate anxiety and depression, the Hospital Anxiety and Depression Scale (HAD) will be used. This scale consists of 14 items, divided into 7 for assessing anxiety and 7 for assessing depression. The items are scored on a rising scale from 0 to 3, with a maximum score of 21 for each subdivision. Higher scores indicate greater levels of anxiety and depression. HADS results are interpreted through scores for anxiety (HADS-A) and depression (HADS-D), with scores ranging from 0 to 21 for each subscale. Higher scores indicate worse depression and anxiety.

OTHER OUTCOMES:
The perceived overall effect - Likert Scale | post eight weeks of intervention.
  To assess the perceived overall effect, the physiotherapist will ask the following question: "Compared to the beginning of the treatment, how would the participant describe your lower back today?" The patient will respond using the Likert Scale. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: KAREN V TRIPPO, PhD, PT, Principal Investigator — Federal University of Bahia
Locations (1):
- Clínica Escola de Fisioterapia da UFBA - CEF/UFBA, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boiko VV, Prasol VA, Peresada II, Karnaukh VF. [Case of successful treatment of gunshot wound of the neck with injury of the carotid artery bifurcation]. Klin Khir. 1995;(7-8):46-7. No abstract available. Russian. PMID 8624945
- [Background] Ferreira GE, Barreto RG, Robinson CC, Plentz RD, Silva MF. Global Postural Reeducation for patients with musculoskeletal conditions: a systematic review of randomized controlled trials. Braz J Phys Ther. 2016 Apr 1;20(3):194-205. doi: 10.1590/bjpt-rbf.2014.0153. PMID 27437710
- [Background] Hisanaga K, Onodera H, Kogure K. Changes in levels of purine and pyrimidine nucleotides during acute hypoxia and recovery in neonatal rat brain. J Neurochem. 1986 Nov;47(5):1344-50. doi: 10.1111/j.1471-4159.1986.tb00763.x. PMID 3020172
- [Background] Johnsn FH, Shimomura O. Preparation and use of aequorin for rapid microdetermination of Ca 2+ in biological systems. Nat New Biol. 1972 Jun 28;237(78):287-8. doi: 10.1038/newbio237287a0. No abstract available. PMID 4402563
- [Background] Cavalcanti IF, Antonino GB, Monte-Silva KKD, Guerino MR, Ferreira APL, das Gracas Rodrigues de Araujo M. Global Postural Re-education in non-specific neck and low back pain treatment: A pilot study. J Back Musculoskelet Rehabil. 2020;33(5):823-828. doi: 10.3233/BMR-181371. PMID 31929138